CLINICAL TRIAL: NCT03576989
Title: Impact of Omega-3 Fatty Acid Oral Therapy on Healing of Chronic Venous Leg Ulcers in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018H0261; R01AG059981 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-07-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Venous Leg Ulcers
Keywords: leg ulcer, fish oil, wounds
MeSH Terms: conditions — Leg Ulcer; Wounds and Injuries | interventions — Eicosapentaenoic Acid; Docosahexaenoic Acids; Fish Oils; Mineral Oil

STUDY DESIGN:
Intervention Model Description: 2-group randomized, double-blind, repeated measures design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators, participants and care providers blinded as to treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPA+DHA Group (Experimental): 12 weeks of daily oral therapy with EPA+DHA (three opaque softgels to provide a total daily intake of 1.87 g of EPA + 1.0 g of DHA)
  Interventions: Dietary Supplement: EPA+DHA
- Placebo Group (Placebo Comparator): 12 weeks of daily oral therapy with placebo (three opaque softgels to provide a total daily intake of 2.5 mL of mineral oil)
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: EPA+DHA — EPA+DHA are the n-3 polyunsaturated fatty acids contained in fish oil
  Other Names: eicosapentaenoic acid + docosahexaenoic acid; fish oil
  Arms: EPA+DHA Group
Other: placebo — placebo contains mineral oil
  Other Names: mineral oil
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to test the efficacy of an oral, nutrient intervention containing the bioactive components of fish oil to promote healing of chronic venous leg ulcers (CVLUs) by reducing the chronic inflammation at wound sites that prevents healing progression. If this systemic, nutrient intervention is found to alter the microenvironment of CVLUs, the science of wound healing and care of patients with CVLUs will be vastly improved.

DETAILED DESCRIPTION:
The pathogenesis of CVLU involves high numbers of activated polymorphonuclear leukocytes (PMN) that are associated with persistent inflammation in the wound bed. The proposed research is to test the efficacy of an oral, nutrient intervention containing the bioactive components of fish oil (eicosapentaenoic acid - EPA + docosahexaenoic acid - DHA) to assuage PMN activity and promote healing. The study plans to include 248 successive eligible adults ≥ 55 years of age with CVLUs who continue to receive standard care at two university out-patient wound clinics. Participants will be randomized to 2 groups: 12 weeks of daily oral therapy with EPA+DHA (1.87 g/d of EPA + 1.0 g/d of DHA) or daily oral therapy with placebo. At 0, 4, 8 and 12 weeks, across the 2 groups, three specific aims will be pursued:

Aim 1. Compare levels of EPA+DHA-derived lipid mediators, and inflammatory cytokines in blood and CVLU fluid.

Subaim 1a. Compare inflammatory cytokine gene expression by PMNs in blood (neutrophils and monocytes).

Aim 2. Compare PMN activation (blood, CVLU fluid), and PMN-derived protease levels (CVLU fluid).

Aim 3. Compare reduction in wound area, controlling for key factors known to affect healing, and determine relationships with lipid mediators, cytokines and PMN activation.

Subaim 3a. Compare frequency of CVLU recurrence and levels of study variables in blood between 2 subgroups within the EPA+DHA group with healed CVLUs (after 3 additional months of EPA+DHA therapy versus placebo therapy beyond Week 12 time point).

Subaim 3b. Compare the symptom of pain at all time points and quality of life at first and last study visits across the 2 groups and 2 subgroups.

ELIGIBILITY:
Inclusion Criteria:

Women and men ≥ 55 years of age with:

* A CVLU between the ankle and knee that has been present for at least 4 weeks, but not longer than 12 months, prescribed compression therapy with 1-4 layer bandaging;
* Ankle brachial pressure index (ABPI) between 0.7 and 1.2;
* Target wound area of 2-60 cm2 who can
* Read and understand English or Spanish, and
* Provide consent.

Exclusion Criteria:

* Fish allergy;
* Corticosteroids or selective cyclooxygenase (COX)-2 inhibitors (e.g., Celebrex); non- steroidal anti-inflammatory drugs (NSAIDS) > 2x/week (exception: aspirin 81 mg/day);
* Autoimmune diseases;
* Chemotherapy within 6 months of Week 0;
* Diabetes if HbA1c > 12% or ulcer complicated by cellulitis, exposed tendon or bone.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Change in EPA+DHA-derived lipid mediators | 0, 4, 8 and 12 weeks
  plasma and wound fluid levels of EPA+DHA-derived lipid mediators of inflammation
Change in inflammatory cytokines | 0, 4, 8 and 12 weeks
  plasma and wound fluid levels of pro- and anti-inflammatory cytokines
Change in polymorphonuclear leukocyte (PMN) activation | 0, 4, 8 and 12 weeks
  blood and wound fluid levels of PMN activation
Change in PMN-derived proteases | 0, 4, 8 and 12 weeks
  wound fluid levels of PMN-derived proteases
Change in reduction in wound area | 0, 4, 8 and 12 weeks
  reduction in wound area measured in cm2

SECONDARY OUTCOMES:
inflammatory cytokine gene expression | 0, 4, 8 and 12 weeks
  inflammatory cytokine gene expression by neutrophils and monocytes from blood
recurrence of chronic venous leg ulcers | 3 months beyond Week 12 time point in participants whose leg ulcers have healed by Week 12
  frequency of recurrence of chronic venous leg ulcers after healing
Change in symptom of pain | 0, 4, 8 and 12 weeks (and at 3 month timepoint beyond Week 12 in participants in extended study - with healed leg ulcers by Week 12)
  pain related to venous leg ulcer measured using the Venous Clinical Severity Score (VCSS)
quality of life using the VEINES-QOL/Sym questionnaire | 0, 12 weeks ((and at 3 month timepoint beyond Week 12 in participants in extended study - with healed leg ulcers by Week 12)
  quality of life related to venous leg ulcer measured using the Venous Insufficiency Epidemiological and Economic Study-Quality of Life/Symptoms questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jodi C McDaniel, PhD, Principal Investigator — Ohio State University, College of Nursing
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McDaniel JC, Rausch J, Tan A. Impact of omega-3 fatty acid oral therapy on healing of chronic venous leg ulcers in older adults: Study protocol for a randomized controlled single-center trial. Trials. 2020 Jan 16;21(1):93. doi: 10.1186/s13063-019-3970-7. PMID 31948466